CLINICAL TRIAL: NCT06764914
Title: NAturheilkundliche Komplextherapie Bei Episodischer MIgräne Und KOpfschmerz Vom Spannungstyp
Brief Title: Integrative and Complementary Therapy for Episodic Migraine and Tension-type Headache
Acronym: NAMIKOS
Status: Not yet recruiting | Type: Observational
Sponsor: Kliniken Essen-Mitte (Other)
Responsible Party: Sponsor
Other Study IDs: 2023273
Record Dates: First submitted 2024-12-12; First posted 2025-01-09 (Actual); Last update posted 2025-01-09 (Actual); Status verified 2025-01

CONDITIONS: Migraine; Headache, Tension-Type
Keywords: Migraine; Headache, Tension-Type
MeSH Terms: conditions — Migraine Disorders; Tension-Type Headache | interventions — Complementary Therapies

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | US Export: No

GROUPS / COHORTS (1):
- episodic migraine and/or episodic tension headache (tension-type headache TTH)
  Interventions: Other: integrative and complementary medicine

INTERVENTIONS:
Other: integrative and complementary medicine — Treatment with integrative and complementary methods for both, inpatients and outpatients, includes conventional therapy, integrative methods and ordinal therapy/MBM, which are individually designed for each patient. Similar to a shedule, with therapy units from the following areas: hydrotherapy/thermotherapy, exercise therapy, physiotherapy, nutritional therapy and bodywork therapy, supplemented as required by phytotherapeutic and other therapies, such as acupuncture, neural therapy and cupping. After inpatient treatment, patients can receive up to 10 additional outpatient treatments at our TCM outpatient clinic. There is also a 10-week programme for day patients. This focuses on ordinal therapy to achieve sustainable, balanced lifestyle changes. This includes classic acupuncture and drainage techniques such as Gua Sha (connective tissue massage in TCM) or cupping, as well as neural therapy, electro-acupuncture and others. Daily medical visits and self-care advice are also included.

SUMMARY:
This study is a monocentric uncontrolled observational study to evaluate a 12-14 day inpatient stay in an internal medicine clinic for integrative and complementary medicine for patients with episodic migraine and/or episodic tension headache. The aim is to investigate the extent to which a 14-day inpatient stay can influence a reduction in headache days and/or pain intensity, medication use, quality of life, anxiety, depression, perceived stress, general well-being, and a reduction in sick days/work absenteeism, and prevent the chronification of migraine and may counteract the chronification of migraine or tension-type headache. In addition, patients' previous experiences with complementary naturopathic therapies, expectations and perceived benefits in everyday life will be analysed.

DETAILED DESCRIPTION:
Primary headache disorders are among the most common neurological disorders worldwide, with a lifetime prevalence of over 90%. Tension-type headache (TTH) is the most common type of primary headache. It manifests as a dull, pressing, tightening pain that usually 'rises' from the neck to the back of the head and down to the temples on both sides, but can theoretically occur in any part of the head. The frequency of pain attacks is used to define episodic (< 15 days/month or < 180 days/year) and chronic TTH (> 15 days/month for > 3 months or > 180 days/year). The main therapeutic options are classical analgesics (non-steroidal anti-inflammatory drugs, NSAIDs; Novalgin) in acute cases or tricyclic antidepressants as prevention. Prophylaxis can be combined with (endurance) exercise or acupuncture. Migraine is rarer than TTH, affecting about 9% of the population, but it is one of the most common causes of disability worldwide. It is defined as a headache with or without preceding neurological symptoms (called an aura) and occurs mainly in middle age, between 20 and 50 years. In acute attacks, migraine headaches are treated with medication (usually classic analgesics such as NSAIDs, Novalgin or migraine-specific triptans). In cases of severe distress due to frequent and severe attacks, medication may also be used as a prophylactic measure. A distinction is also made between episodic migraine (< 15 days in the last 3 months) and chronic migraine (> 15 days/month in the last 3 months). In addition to drug therapy there are also non-drug approaches such as acupuncture, behavioural therapy, biofeedback or relaxation techniques, which may be combined with drug prophylaxis. Complications of migraine include status migraenosus (migraine attacks lasting more than 72 hours), migraine stroke and/or chronicisation of migraine. The headache disorders listed above can occur alone or in combination. When they occur together, they can severely restrict a person's daily life. According to the German Society of Neurology (DGN-Deutsche Gesellschaft für Neurologie), multimodal approaches, such as inpatient multimodal pain therapy, are explicitly recommended only in the context of chronic headache, especially chronic migraine. In addition, there are often life-limiting comorbidities, which often worsen with chronicity. The Clinic for Integrative and Complementary Medicine at the Evangelische Kliniken Essen-Mitte has been treating patients with various pain disorders for more than 20 years. Within the framework of so-called integrative care concepts with the Techniker Krankenkasse (TK) and the Barmer Ersatzkasse (BEK), headache patients are treated with naturopathic-integrative methods both as inpatients and as outpatients. The aim of this prospective observational study is to evaluate the integrative-complementary concept in patients with episodic headache (migraine and/or tension headache) without medication abuse or medication-induced headache. It will be observed whether this concept can reduce sick days/work absences, pain intensity and frequency, and medication use, thus preventing chronicity.

ELIGIBILITY:
Inclusion Criteria:

* Episodic migraine (<15 headache days/month in the last 3 months)
* Episodic tension headache (<15 headache days/month in the last 3 months)
* Mixed forms or parallel occurrence of both types of headache is permitted
* Diagnosis confirmed in advance by a neurologist
* Mandatory imaging to exclude another cause of headache before or during hospitalisation (cMRI or cCT)
* Participation in the integrative headache supply programm oft the health insurence provider Barmer Ersatzkasse and Techniker Krankenkasse
* Signed declaration of consent

Exclusion Criteria:

* Age younger than 18 years
* Chronic migraine (15 migraine days in the last 3 months) or chronic tension type headache
* Medication-induced headache/painkiller abuse (> 10 triptans/combination analgesics/ergotamines/opiates or >15 classical analgesics per month)
* Acute severe mental illness (e.g. severe depression with suicidal tendencies)
* Acute, severe physical illness that prevents participation in the inpatient naturopathic programme or emergency inpatient treatment of a different kind (e.g. ongoing treatment of a cancer severe acute illness of the cardiovascular system such as heart attack, stroke, acute insufficiency of other organs (kidney, liver, etc.), other severe acute neurological diseases, e.g. relapse of multiple sclerosis, uncontrolled epilepsy)
* Pregnancy/lactation period
* Simultaneous participation in other clinical studies
* No consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with episodic headaches (TTH and/or migraine) who choose to spend 12 to 14 days at the Clinic for Integrative and Complementary Medicine. The diagnosis must be confirmed by a neurological examination.
Sampling Method: Non-Probability Sample
Enrollment: 130 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2030-01-01 (Estimated); Study Completion 2031-01-01 (Estimated)

PRIMARY OUTCOMES:
Number of headache days/month (headache diary); | 48 weeks after inpatient hospitalisation

SECONDARY OUTCOMES:
Pain Perception Scale (PPS) using a visual analogue scale (VAS) | 48 weeks after inpatient hospitalisation
  The Pain Perception Scale is a tool to measure the patient's subjective assessment of symptoms, using the visual analogue scale of pain intensity to record pain on a scale from '0' to '10'. '0' is no pain and '10' is the highest level of pain.
Number of sick days from T0 to T3 (headache diary) | 48 weeks after inpatient hospitalisation
- Number of painkillers/month (headache diary) | 48 weeks after inpatient hospitalisation
Headache Disability Index (HDI) | 48 weeks after inpatient hospitalisation
  HDI measure the impact of headache disorders on quality of life. The HDI is a 27-item questionnaire. The first two questions relate to frequency (once per month; more than once per month but less than four per month; more than once per week) and intensity ('mild', 'moderate' and 'severe').
  The remaining 25 questions are designed to assess the quality of life affected by headache. Each question can be scored from 0 to 4 points. A total score of '10-28' indicates mild disability, '30-48' is moderate, '50-68' is severe and '72' or more is complete disability.
Short-Form Health Survey (SF-12) | 48 weeks after inpatient hospitalisation
  The Short-Form Health Survey 12 assesses the impact of health on an individual's daily life. The SF-12 theoretically ranges from '0' (lowest possible quality of life) to '100' (highest possible quality of life). The SF-12 measures disease-related quality of life using 12 items divided into 8 subscales. Higher scores indicate better quality of life.
Hospital Anxiety and Depression Scale (HADS) | 48 weeks after inpatient hospitalisation
  Anxiety and depression are measured using the HADS. The questionnaire contains 14 items, 7 on the anxiety scale and 7 on the depression scale. Total scores on the HADS-A (anxiety) and HADS-D (depression) scales range from '0-21', with higher scores indicating higher levels of anxiety/depression. Scores of '0-7' per HADS subscale (HADS-A/D) are considered 'normal', '8-10' as 'mild', scores above '11' as severe (up to '14' 'moderate', '15-21' 'severe').
Flourishing Scale (FS) | 48 weeks after inpatient hospitalisation
  Subjective well-being is assessed using the Flourishing Scale. This consists of 8 socio-psychological well-being items that can be scored on a scale from '1' to '7'. The possible range of the total score is from '8' (lowest possible score) to '56' (highest possible score). A high score corresponds to a person with many psychological resources and strengths.
Perception Stress Scale (PSS-10) | 48 weeks after inpatient hospitalisation
  Perceived stress is measured using two scales (helplessness and self-efficacy) based on 10 items. The scales can be scored from '0' (never) to '5' (very often). The total score is calculated as the sum of the helplessness scale items and the sum of the inverted self-efficacy scale items. Higher scores indicate higher levels of stress.

OTHER OUTCOMES:
- Causation and Intensity of Adverse events (AEs) | 12 months after inpatient hospitalisation
  negative side effects
Medical service use figures | 48 weeks after inpatient hospitalisation
  Previous experience, use and expectations of integrative and complementary therapies will also be assessed using socio-demographic data.
Work ability | 48 weeks after inpatient hospitalisation
  Work ability is recorded as part of the socio-demographic data and can be rated on a scale from '0' (total inability to work) to '10' (best possible ability to work).

CONTACTS AND LOCATIONS:
Overall Officials: Petra Voiß, PD Dr. med., Study Chair — Evang. Kliniken Essen-Mitte, Clinic for Integrative Oncology & Supportivemedicine